CLINICAL TRIAL: NCT02034006
Title: A 12-month, Open-label, Interventional, Multicentre Study to Investigate the Current Criteria Driving Re-treatment With Ranibizumab Upon Relapse in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia
Brief Title: A Study of the Criteria Establishing the Need for Re-treatment With Ranibizumab Upon Relapse in Patients With Visual Impairment Due to Choroidal Neovascularization Secondary to Pathologic Myopia.
Acronym: OLIMPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002FIT01; 2013-003334-33 (EudraCT Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-10

CONDITIONS: Choroidal Neovascularization Secondary to Pathologic Myopia
Keywords: pathological myopia; choroidal neovascularization; ranibizumab; mono-bilateral; poor visual acuity; retinal disease; eye disease; Angiogenesis Inhibitors; Angiogenesis Modulating Agents
MeSH Terms: conditions — Myopia, Degenerative; Choroidal Neovascularization; Retinal Diseases; Eye Diseases | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ranibizumab (Experimental): Patients treated with a single ranibizumab 0.5 mg/0.05ml intravitreal injection
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — All patients received a single initial intravitreal injection of ranibizumab 0.5 mg/0.05 ml as per Committee for Human Medicinal Products (CHMP)approval. Further injections might have been required when monitoring reveals disease activity. Disease activity, defined as reduced visual acuity and/or signs of lesion activity, was evaluated based on clinical examination (BCVA, fundus), and/or optical coherence tomography (OCT), and/or fluorescein angiography (FAG). Bilateral treatment was allowed provided at least 14 days of intercurrence.
  Other Names: RFB002

SUMMARY:
The primary objective of the study was to investigate current criteria driving re-treatment in patients affected by Choroidal Neovascularization (CNV) secondary to Pathologic Myopia (PM) and experiencing a relapse of the disease after the first administration of ranibizumab.

ELIGIBILITY:
INCLUSION CRITERIA:

* Written informed consent given before any study related procedure is performed
* Diagnosis of active CNV secondary to PM confirmed by complete ocular examination in the affected eye(s) using the following criteria:
* Presence of high myopia greater than -6D of spherical equivalence
* Presence of posterior changes compatible with pathologic myopia (any signs of attenuation of retinal pigment epithelium (RPE) and choroids, mottling of the RPE, tilted disc, geographic atrophy of RPE, Fuchs spots, posterior staphyloma, submacular hemorrhage, lacquer cracks) detected by fundus ophthalmoscopy and fundus photography
* Presence of active leakage from CNV observed through fluorescein angiography (FAG)
* Presence of intra or subretinal fluid demonstrated by Optical Coherence Tomography (OCT)
* BCVA > 24 letters and < 78 letters tested at 4 meters staring distance using ETDRS-like visual acuity chart
* Visual loss must be only due to the presence of any eligible types of CNV related to PM based on clinical ocular findings, FAG and OCT. (Also patients that have for example 20/60 as their best visual acuity due to PM in their history and have additional vision loss due to CNV lesion can be included)

EXCLUSION CRITERIA:

* Patients with inability to comply with study related procedures
* Pregnant or nursing (lactating) women and women of childbearing potential UNLESS using effective contraception during treatment
* Presence of confirmed systolic blood pressure > 150 mmHg or diastolic > 90 mmHg at the time of enrollment
* History of stroke
* Any type of advanced, severe or unstable medical condition or its treatment that could significantly bias the assessment of clinical status and interfere with primary and/or secondary outcome evaluations or put the patient at risk
* Presence of active infectious disease or intra-ocular inflammation in either eye at the time of enrollment
* Ocular disorders in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 12-month study period (including retinal detachment, cataract and pre-retinal membrane of the macula)
* History of pan-retinal or focal/grid laser photocoagulation with involvement of the macular area in the study eye at any time
* History of intraocular treatment with any anti-vascular endothelial growth factor (VEGF), verteporfin photodynamic therapy (vPDT) and any intra-ocular surgery or corticosteroid administration within one month before study entrance
* Known hypersensitivity to ranibizumab or any component of the ranibizumab formulation
* Simultaneous participation in a study that includes administration of any investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Italy (25):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Desenzano del Garda, BS
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rapallo, GE
  - Novartis Investigative Site, Terracina, LT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Conegliano, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli

REFERENCES:
- [Derived] Ricci F, Staurenghi G, Varano M, Eandi C, Sinibaldi TL, Colombo L, Bartezaghi M, Bassanini S. OLIMPIC: a 12-month study on the criteria driving retreatment with ranibizumab in patients with visual impairment due to myopic choroidal neovascularization. Graefes Arch Clin Exp Ophthalmol. 2019 Apr;257(4):759-768. doi: 10.1007/s00417-019-04248-8. Epub 2019 Jan 24. PMID 30680452

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred fifteen (215) subjects were screened in this study (i.e. provided written informed consent). Two hundred (200) subjects underwent baseline visit and received at least one injection of ranibizumab.
Groups:
- Ranibizumab: All subjects who received at least one dose of ranibizumab
Period: Overall Study
Arm/Group | Ranibizumab
Started | 200
Once Treated Patients | 70
Re-treated Patients | 130
Completed | 186
Not Completed | 14
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 5
Not completed — Death | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All subjects who received at least one dose of ranibizumab
Groups:
- Ranibizumab: Treated Once: Patients treated only once with a single ranibizumab 0.5 mg/0.05ml intravitreal injection.
- Ranibizumab: Re-treated Once: Patients treated more than once with a single ranibizumab 0.5 mg/0.05ml intravitreal injection.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once | Total
Number analyzed (Participants) | 70 | 130 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.27 (13.03) | 62.12 (12.52) | 61.82 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 94 | 147
  Male | 17 | 36 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Active Leakage
Description: Presence of active leakage on fluorescein angiography (FAG) was assessed at screening (14 to 3 days before baseline visit), month 2 and month 6. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of presence of active leakage (Yes/No). For retreated patients, the presence/absence of active leakage was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis. *NE = Not evaluable
Time Frame: Screening, Month 2, Month 6
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and underwent fluorescein angiography at that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Screening: Active leakage, No: number analyzed (Participants) | 64 | 124
  Screening: Active leakage, No | 3 | 0
  Screening: Active leakage, Yes: number analyzed (Participants) | 64 | 124
  Screening: Active leakage, Yes | 61 | 121
  Screening: Active leakage, NE: number analyzed (Participants) | 64 | 124
  Screening: Active leakage, NE | 0 | 2
  Screening: Active leakage, Missing: number analyzed (Participants) | 64 | 124
  Screening: Active leakage, Missing | 0 | 1
  Month 2: Active leakage, No: number analyzed (Participants) | 61 | 119
  Month 2: Active leakage, No | 58 | 61
  Month 2: Active leakage, Yes: number analyzed (Participants) | 61 | 119
  Month 2: Active leakage, Yes | 3 | 56
  Month 2: Active leakage, NE: number analyzed (Participants) | 61 | 119
  Month 2: Active leakage, NE | 0 | 2
  Month 6: Active leakage, No: number analyzed (Participants) | 60 | 115
  Month 6: Active leakage, No | 55 | 73
  Month 6: Active leakage, Yes: number analyzed (Participants) | 60 | 115
  Month 6: Active leakage, Yes | 4 | 40
  Month 6: Active leakage, NE: number analyzed (Participants) | 60 | 115
  Month 6: Active leakage, NE | 1 | 2
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Presence vs. absence of active leakage; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 72.37, 95% CI 2-sided [23.44 to 223.42]

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Baseline to Month 6 and Month 12 on Study Eye
Description: Change from baseline in BCVA (Best Corrected Visual Acuity) was Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score. Patients with a BCVA ETDRS letter score of 78 to 24 in the study eye were included; A higher score represents better functioning of the study eye. A positive change from baseline shows improvement.
Time Frame: Baseline, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab. The study eyes of the patients belonging to the FAS were analyzed.
Measure: Mean (Standard Deviation); unit: letters
Units Other Than Participants: study eyes
Groups:
- Ranibizumab: Patients treated with a single ranibizumab 0.5 mg/0.05ml intravitreal injection. Further injections might be required when monitoring reveals disease activity.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 200
Number analyzed (study eyes) | 200
letters
  Change at 6 month: number analyzed (study eyes) | 190
  Change at 6 month | 7.51 (11.68)
  Change at 12 month: number analyzed (study eyes) | 191
  Change at 12 month | 8.42 (12.81)

3. Secondary Outcome: Mean Number of Ranibizumab Injection
Description: Mean number of ranibizumab injection is reported as number of injections per patient.
Time Frame: Baseline to Month 12
Population: Full Analysis Set (FAS): all subjects who received at least one dose of ranibizumab
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Ranibizumab
Number analyzed (Participants) | 200
injections | 2.41 (1.53)

4. Secondary Outcome: Time to Re-treatment
Description: Time to re-treatment, defined as time in months from the data of first dose of ranibizumab to the date of re-treatment, was evaluated.
Time Frame: Baseline to Month 12
Population: Full Analysis Set (FAS): all subjects who received at least one dose of ranibizumab
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 130
Months | 2.56 (2.17)

5. Secondary Outcome: Number of Patients Having Ocular and/or Systemic Adverse Event (AE)
Description: Number of patients with any systemic AE, with serious systemic AE, with an ocular AE, with an ocular serious AE are reported
Time Frame: Baseline to Month 12
Population: Safety Population: all subjects who received at least one dose of ranibizumab and had at least one post-baseline safety assessment.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab
Number analyzed (Participants) | 200
Patients
  Any systemic Adverse Event | 30
  Serious systemic Adverse Event | 5
  Ocular Adverse Event | 41
  Ocular serious adverse event | 2

6. Secondary Outcome: Change in Patient Quality of Life From Baseline to Month 2 and Month 12
Description: Patient quality of life was assessed by Impact of Vision Impairment (IVI) questionnaire. IVI is a 32-item instrument, either self- or interviewer-administered, developed to measure the impact of vision impairment on daily activities in five domains. The 32 items were divided into 5 domains as follows: Leisure and work (items 1 to 5), Social and consumer interaction (items 6 to 10 and items 23-24), Household and personal care (items 11 to 14 and items 20-21), Mobility (items 15 to 19 and item 22), Emotional reaction to vision loss (items 25 to 32). Responses to the IVI items were rated on a five-category Likert scale: not at all, 0; hardly at all, 1; a little, 2; a fair amount, 3; a lot, 4; and can't do because of eyesight, 5. Total score was an arithmetic average of the items rated between 0 (the best score) and 5 (the worst score). A negative change indicates improvement. Data was computed on items with non missing response
Time Frame: Baseline, Month 2, Month 12
Population: Full Analysis Set (FAS): all subjects who received at least one dose of ranibizumab with data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
units on a scale
  Change at Month 2: number analyzed (Participants) | 60 | 124
  Change at Month 2 | -0.40 (0.68) | -0.15 (0.60)
  Change at month 12: number analyzed (Participants) | 59 | 122
  Change at month 12 | -0.54 (0.91) | -0.36 (0.81)

7. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Macular Edema
Description: Presence of macular edema from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of presence of macular edema (Yes/No). For retreated patients, the presence/absence of macular edema was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis. *NE = Not evaluable
Time Frame: Screening, Month 2, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and underwent OCT at that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Screening: Macular Edema, No: number analyzed (Participants) | 69 | 129
  Screening: Macular Edema, No | 38 | 63
  Screening: Macular Edema, Yes: number analyzed (Participants) | 69 | 129
  Screening: Macular Edema, Yes | 28 | 65
  Screening: Macular Edema, NE: number analyzed (Participants) | 69 | 129
  Screening: Macular Edema, NE | 3 | 1
  Month 2: Macular Edema, No: number analyzed (Participants) | 69 | 129
  Month 2: Macular Edema, No | 59 | 103
  Month 2: Macular Edema, Yes: number analyzed (Participants) | 63 | 129
  Month 2: Macular Edema, Yes | 3 | 24
  Month 2: Macular Edema, NE: number analyzed (Participants) | 63 | 129
  Month 2: Macular Edema, NE | 1 | 2
  Month 6: Macular Edema, No: number analyzed (Participants) | 60 | 126
  Month 6: Macular Edema, No | 57 | 101
  Month 6: Macular Edema, Yes: number analyzed (Participants) | 60 | 126
  Month 6: Macular Edema, Yes | 2 | 24
  Month 6: Macular Edema, NE: number analyzed (Participants) | 60 | 126
  Month 6: Macular Edema, NE | 1 | 1
  Month 12: Macular Edema, No: number analyzed (Participants) | 61 | 124
  Month 12: Macular Edema, No | 56 | 108
  Month 12: Macular Edema, Yes: number analyzed (Participants) | 61 | 124
  Month 12: Macular Edema, Yes | 4 | 15
  Month 12: Macular Edema, NE: number analyzed (Participants) | 61 | 124
  Month 12: Macular Edema, NE | 1 | 1
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Presence vs. absence of macular edema; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 9.33, 95% CI 2-sided [3.18 to 27.36]

8. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Cysts
Description: Presence of cysts from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of presence of cysts (Yes/No). For retreated patients, the presence/absence of cysts was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis. *NE = Not evaluable
Time Frame: Screening, Month 2, Month 6, Month 12
Population: as for outcome 7
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Screening: Cysts, No: number analyzed (Participants) | 69 | 129
  Screening: Cysts, No | 41 | 79
  Screening: Cysts, Yes: number analyzed (Participants) | 69 | 129
  Screening: Cysts, Yes | 27 | 50
  Screening: Cysts, NE: number analyzed (Participants) | 69 | 129
  Screening: Cysts, NE | 1 | 0
  Month 2: Cysts, No: number analyzed (Participants) | 63 | 129
  Month 2: Cysts, No | 60 | 94
  Month 2: Cysts, Yes: number analyzed (Participants) | 63 | 129
  Month 2: Cysts, Yes | 2 | 32
  Month 2: Cysts, NE: number analyzed (Participants) | 63 | 129
  Month 2: Cysts, NE | 1 | 2
  Month 2: Cysts, Missing: number analyzed (Participants) | 63 | 129
  Month 2: Cysts, Missing | 0 | 1
  Month 6: Cysts, No: number analyzed (Participants) | 60 | 126
  Month 6: Cysts, No | 57 | 98
  Month 6: Cysts, Yes: number analyzed (Participants) | 60 | 126
  Month 6: Cysts, Yes | 2 | 27
  Month 6: Cysts, NE: number analyzed (Participants) | 60 | 126
  Month 6: Cysts, NE | 1 | 1
  Month 12: Cysts, No: number analyzed (Participants) | 61 | 124
  Month 12: Cysts, No | 57 | 97
  Month 12: Cysts, Yes: number analyzed (Participants) | 61 | 124
  Month 12: Cysts, Yes | 3 | 26
  Month 12: Cysts, NE: number analyzed (Participants) | 61 | 124
  Month 12: Cysts, NE | 1 | 1
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Presence vs. absence of cysts; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 12.66, 95% CI 2-sided [3.76 to 42.67]

9. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Intra-retinal Fluid
Description: Presence of Intra-retinal fluid from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of presence of Intra-retinal fluid (Yes/No). For retreated patients, the presence/absence of Intra-retinal fluid was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis. *NE = Not evaluable
Time Frame: Screening, Month 2, Month 6, Month 12
Population: as for outcome 7
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Screening: Intra-retinal fluid, No: number analyzed (Participants) | 69 | 129
  Screening: Intra-retinal fluid, No | 19 | 37
  Screening: Intra-retinal fluid, Yes: number analyzed (Participants) | 69 | 130
  Screening: Intra-retinal fluid, Yes | 49 | 90
  Screening: Intra-retinal fluid, NE: number analyzed (Participants) | 69 | 129
  Screening: Intra-retinal fluid, NE | 1 | 2
  Month 2: Intra-retinal fluid, No: number analyzed (Participants) | 63 | 129
  Month 2: Intra-retinal fluid, No | 55 | 77
  Month 2: Intra-retinal fluid, Yes: number analyzed (Participants) | 63 | 129
  Month 2: Intra-retinal fluid, Yes | 7 | 50
  Month 2: Intra-retinal fluid, NE: number analyzed (Participants) | 63 | 129
  Month 2: Intra-retinal fluid, NE | 1 | 2
  Month 6: Intra-retinal fluid, No: number analyzed (Participants) | 60 | 130
  Month 6: Intra-retinal fluid, No | 57 | 85
  Month 6: Intra-retinal fluid, Yes: number analyzed (Participants) | 60 | 126
  Month 6: Intra-retinal fluid, Yes | 1 | 38
  Month 6: Intra-retinal fluid, NE: number analyzed (Participants) | 60 | 126
  Month 6: Intra-retinal fluid, NE | 2 | 3
  Month 12: Intra-retinal fluid, No: number analyzed (Participants) | 61 | 124
  Month 12: Intra-retinal fluid, No | 58 | 96
  Month 12: Intra-retinal fluid, Yes: number analyzed (Participants) | 61 | 124
  Month 12: Intra-retinal fluid, Yes | 2 | 26
  Month 12: Intra-retinal fluid, NE: number analyzed (Participants) | 61 | 124
  Month 12: Intra-retinal fluid, NE | 1 | 2
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Presence vs. absence of intra-retinal fluid; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 49.80, 95% CI 2-sided [11.62 to 213.50]

10. Primary Outcome: Change in Central Subfield Thickness (CSFT)
Description: Central subfield thickness (CSFT) from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of change in CSFT versus previous visit. For retreated patients, the change in CSFT was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Screening, Month 2, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and underwent OCT at that time point and previous visit.
Measure: Mean (Standard Deviation); unit: micromilimeter(um)
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
micromilimeter(um)
  Month 2 Vs. Screening : CSFT: number analyzed (Participants) | 61 | 125
  Month 2 Vs. Screening : CSFT | -16.15 (86.65) | -34.28 (78.01)
  Month 6 Vs. Month 2: CSFT: number analyzed (Participants) | 57 | 121
  Month 6 Vs. Month 2: CSFT | -11.04 (61.06) | -15.83 (70.74)
  Month 12 Vs. Month 6: CSFT: number analyzed (Participants) | 57 | 119
  Month 12 Vs. Month 6: CSFT | 1.29 (62.55) | 8.64 (76.79)
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Change in Central subfield thickness vs previous visit; Test type: Superiority or Other; p = 0.1514, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.99 to 1.00]

11. Primary Outcome: Change in Central Subfield Volume (CSV)
Description: Central subfield volume (CSV) from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of change in CSV versus previous visit. For retreated patients, the change in CSV was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Screening, Month 2, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and underwent OCT at that time point and the previous visit.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
mm^3
  Month 2 Vs. Screening : CSV: number analyzed (Participants) | 49 | 96
  Month 2 Vs. Screening : CSV | -0.02 (0.06) | -0.02 (0.06)
  Month 6 Vs. Month 2: CSV: number analyzed (Participants) | 48 | 97
  Month 6 Vs. Month 2: CSV | -0.00 (0.04) | -0.01 (0.07)
  Month 12 Vs. Month 6: CSV: number analyzed (Participants) | 49 | 101
  Month 12 Vs. Month 6: CSV | -0.00 (0.04) | 0.01 (0.08)
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Change in Central subfield volume vs previous visit; Test type: Superiority or Other; p = 0.1265, Regression, Logistic; Odds Ratio (OR) = 0.00, 95% CI 2-sided [0.00 to 5.63]

12. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Sub-retinal Fluid
Description: Presence of sub-retinal fluid from optical coherence tomography (OCT) was assessed at screening (14 to 3 days before baseline visit), month 2, month 6 and month 12. The regression model for sub-retinal fluid was not valid because "Yes" was reported in almost all subjects causing a quasi-complete separation of data points. *NE = Not evaluable
Time Frame: Screening, Month 2, Month 6, Month 12
Population: as for outcome 7
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Screening: Sub-retinal fluid, No: number analyzed (Participants) | 69 | 129
  Screening: Sub-retinal fluid, No | 43 | 65
  Screening: Sub-retinal fluid, Yes: number analyzed (Participants) | 69 | 129
  Screening: Sub-retinal fluid, Yes | 25 | 61
  Screening: Sub-retinal fluid, NE: number analyzed (Participants) | 69 | 129
  Screening: Sub-retinal fluid, NE | 1 | 3
  Month 2: Sub-retinal fluid, No: number analyzed (Participants) | 63 | 130
  Month 2: Sub-retinal fluid, No | 58 | 108
  Month 2: Sub-retinal fluid, Yes: number analyzed (Participants) | 63 | 129
  Month 2: Sub-retinal fluid, Yes | 2 | 17
  Month 2: Sub-retinal fluid, NE: number analyzed (Participants) | 63 | 129
  Month 2: Sub-retinal fluid, NE | 3 | 4
  Month 6: Sub-retinal fluid, No: number analyzed (Participants) | 60 | 126
  Month 6: Sub-retinal fluid, No | 58 | 109
  Month 6: Sub-retinal fluid, Yes: number analyzed (Participants) | 60 | 126
  Month 6: Sub-retinal fluid, Yes | 0 | 14
  Month 6: Sub-retinal fluid, NE: number analyzed (Participants) | 60 | 126
  Month 6: Sub-retinal fluid, NE | 2 | 3
  Month 12: Sub-retinal fluid, No: number analyzed (Participants) | 61 | 124
  Month 12: Sub-retinal fluid, No | 60 | 113
  Month 12: Sub-retinal fluid, Yes: number analyzed (Participants) | 61 | 124
  Month 12: Sub-retinal fluid, Yes | 0 | 8
  Month 12: Sub-retinal fluid, NE: number analyzed (Participants) | 61 | 124
  Month 12: Sub-retinal fluid, NE | 1 | 3

13. Primary Outcome: Number of Patients Treated and Re-treated Based on Presence/Absence of Clinically Significant Abnormalities
Description: Presence of clinically significant abnormalities was assessed at baseline, month 1, month 2, month 3, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of presence of clinically significant abnormalities (Yes/No). For retreated patients, the presence/absence of clinically significant abnormalities was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and underwent ocular examination during that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Baseline: Clinically Significant Abnormal, No | 61 | 103
  Baseline: Clinically Significant Abnormal, Yes | 9 | 27
  Baseline: Clinically Significant Abnormal, Missing | 0 | 0
  Month 1: Clinically Significant Abnorma, No | 60 | 106
  Month 1: Clinically Significant Abnormal, Yes | 6 | 24
  Month 1: Clinically Significant Abnormal, Missing | 4 | 0
  Month 2: Clinically Significant Abnormal, No | 60 | 103
  Month 2: Clinically Significant Abnormal, Yes | 5 | 26
  Month 2:Clinically Significant Abnormal, Missing | 5 | 1
  Month 3: Clinically Significant Abnormal, No | 56 | 108
  Month 3: Clinically Significant Abnormal, Yes | 7 | 20
  Month 3: Clinically Significant Abnormal, Missing | 7 | 2
  Month 6: Clinically Significant Abnormal, No | 59 | 110
  Month 6: Clinically Significant Abnormal, Yes | 3 | 18
  Month 6: Clinically Significant Abnormal, Missing | 8 | 2
  Month 12: Clinically Significant Abnormal, No | 61 | 116
  Month 12: Clinically Significant Abnormal, Yes | 2 | 12
  Month 12: Clinically Significant Abnormal, Missing | 7 | 2
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Presence vs. absence of clinically significant abnormalities; Test type: Superiority or Other; p = 0.0103, Regression, Logistic; Odds Ratio (OR) = 6.91, 95% CI 2-sided [1.58 to 30.23]

14. Primary Outcome: Number of Patients Treated and Re-treated Based on Improvement in Best Corrective Visual Acuity (BCVA) < 5 Letters
Description: Improvement in BCVA < 5 letters (Yes/No) was assessed at month1, month 2, month 3, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of improvement in BCVA < 5 letters (Yes/No) which was reported as Gain >= 5 letters versus Gain < 5 letters. For retreated patients, Gain >= 5 letters and Gain < 5 letters were considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab with improvement in BCVA < 5 letters from baseline at that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Month 1: Gain >= 5 letters: number analyzed (Participants) | 51 | 97
  Month 1: Gain >= 5 letters | 37 | 69
  Month 1: Gain < 5 letters: number analyzed (Participants) | 51 | 97
  Month 1: Gain < 5 letters | 14 | 28
  Month 2: Gain >= 5 letters: number analyzed (Participants) | 50 | 95
  Month 2: Gain >= 5 letters | 38 | 70
  Month 2: Gain < 5 letters: number analyzed (Participants) | 50 | 95
  Month 2: Gain < 5 letters | 12 | 25
  Month 3: Gain >= 5 letters: number analyzed (Participants) | 52 | 94
  Month 3: Gain >= 5 letters | 37 | 74
  Month 3: Gain < 5 letters: number analyzed (Participants) | 52 | 94
  Month 3: Gain < 5 letters | 15 | 20
  Month 6: Gain >= 5 letters: number analyzed (Participants) | 48 | 92
  Month 6: Gain >= 5 letters | 40 | 70
  Month 6: Gain < 5 letters: number analyzed (Participants) | 48 | 92
  Month 6: Gain < 5 letters | 8 | 22
  Month 12: Gain >= 5 letters: number analyzed (Participants) | 51 | 92
  Month 12: Gain >= 5 letters | 43 | 69
  Month 12: Gain < 5 letters: number analyzed (Participants) | 51 | 92
  Month 12: Gain < 5 letters | 8 | 23
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Gain < 5 letters vs. Gain >= 5 letters; Test type: Superiority or Other; p = 0.0854, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.90 to 5.33]

15. Primary Outcome: Number of Patients Treated and Re-treated Based on Improvement in Best Corrective Visual Acuity (BCVA) < 10 Letters
Description: Improvement in BCVA < 10 letters (Yes/No) was assessed at month1, month 2, month 3, month 6 and month 12. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of improvement in BCVA < 10 letters (Yes/No) which was reported as Gain >= 10 letters versus Gain < 10 letters. For retreated patients, Gain >= 10 letters and Gain < 10 letters were considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab with improvement in BCVA < 10 letters from baseline to that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Month 1: Gain >= 10 letters: number analyzed (Participants) | 51 | 97
  Month 1: Gain >= 10 letters | 13 | 27
  Month 1: Gain < 10 letters: number analyzed (Participants) | 51 | 97
  Month 1: Gain < 10 letters | 38 | 70
  Month 2: Gain >= 10 letters: number analyzed (Participants) | 50 | 95
  Month 2: Gain >= 10 letters | 20 | 40
  Month 2: Gain < 10 letters: number analyzed (Participants) | 50 | 95
  Month 2: Gain < 10 letters | 30 | 55
  Month 3: Gain >= 10 letters: number analyzed (Participants) | 52 | 94
  Month 3: Gain >= 10 letters | 22 | 41
  Month 3: Gain < 10 letters: number analyzed (Participants) | 52 | 94
  Month 3: Gain < 10 letters | 30 | 53
  Month 6: Gain >= 10 letters: number analyzed (Participants) | 48 | 92
  Month 6: Gain >= 10 letters | 29 | 50
  Month 6: Gain < 10 letters: number analyzed (Participants) | 48 | 92
  Month 6: Gain < 10 letters | 19 | 42
  Month 12: Gain >= 10 letters: number analyzed (Participants) | 51 | 92
  Month 12: Gain >= 10 letters | 28 | 48
  Month 12: Gain < 10 letters: number analyzed (Participants) | 51 | 92
  Month 12: Gain < 10 letters | 23 | 44
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Gain < 10 letters vs. Gain >= 10 letters; Test type: Superiority or Other; p = 0.0114, Regression, Logistic; Odds Ratio (OR) = 2.52, 95% CI 2-sided [1.23 to 5.17]

16. Primary Outcome: Number of Patients in Different Categories of Changes From Baseline in BCVA
Description: Changes from baseline in BCVA are described for the ETDRS parameter considering the following categories at each assessment: "no change" if the change was equal to 0 letter, "worsening" if change < 0 letter , "improvement" if change > 0 letter. A univariate logistic regression model was applied expressing the presence/absence of the first retreatment in function of change from baseline in BCVA (improved/worsened/stable) which was reported as Improved versus no change and worsened versus no change. For retreated patients, this variable was considered at the closest time-point to the first re-treatment: the last scheduled assessment immediately before the first re-treatment was considered. For treated patients, the last scheduled assessment available was considered. In case of missing value on the scheduled assessment, the value was considered as missing for this analysis.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 6, Month 12
Population: Full Analysis Set (FAS): all patients who received at least one dose of ranibizumab and evaluable BCVA at baseline and that time point.
Measure: Number; unit: Patients
Arm/Group | Ranibizumab: Treated Once | Ranibizumab: Re-treated Once
Number analyzed (Participants) | 70 | 130
Patients
  Month 1: No change: number analyzed (Participants) | 66 | 130
  Month 1: No change | 7 | 18
  Month 1: Worsening: number analyzed (Participants) | 66 | 130
  Month 1: Worsening | 8 | 15
  Month 1: Improvement: number analyzed (Participants) | 66 | 130
  Month 1: Improvement | 51 | 97
  Month 2: No change: number analyzed (Participants) | 65 | 129
  Month 2: No change | 6 | 9
  Month 2: Worsening: number analyzed (Participants) | 65 | 129
  Month 2: Worsening | 9 | 25
  Month 2: Improvement: number analyzed (Participants) | 65 | 129
  Month 2: Improvement | 50 | 95
  Month 3: No change: number analyzed (Participants) | 63 | 128
  Month 3: No change | 3 | 9
  Month 3: Worsening: number analyzed (Participants) | 63 | 128
  Month 3: Worsening | 8 | 25
  Month 3: Improvement: number analyzed (Participants) | 63 | 128
  Month 3: Improvement | 52 | 94
  Month 6: No change: number analyzed (Participants) | 62 | 128
  Month 6: No change | 5 | 6
  Month 6: Worsening: number analyzed (Participants) | 62 | 128
  Month 6: Worsening | 9 | 30
  Month 6: Improvement: number analyzed (Participants) | 62 | 128
  Month 6: Improvement | 48 | 92
  Month 12: No change: number analyzed (Participants) | 63 | 128
  Month 12: No change | 3 | 7
  Month 12: Worsening: number analyzed (Participants) | 63 | 128
  Month 12: Worsening | 9 | 29
  Month 12: Improvement: number analyzed (Participants) | 63 | 128
  Month 12: Improvement | 51 | 92
Statistical Analysis 1: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Change from baseline in BCVA: Improved vs. No change. For retreated subjects, the last scheduled assessment prior to the first retreatment was considered. For subjects treated only once, the last scheduled assessment available was considered; Test type: Superiority or Other; p = 0.0049, Regression, Logistic; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.25 to 0.91]
Statistical Analysis 2: Comparison: Ranibizumab: Treated Once vs Ranibizumab: Re-treated Once; Change from baseline in BCVA: Worsened vs. No change; Test type: Superiority or Other; p = 0.0461, Regression, Logistic; Odds Ratio (OR) = 5.53, 95% CI 2-sided [0.69 to 44.52]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of treatment until exit from the study (approximately 12 months)
Description: Safety Population: All subjects who received at least one dose of ranibizumab and had at least one post-baseline safety assessment.
Groups:
- Ranibizumab: All subjects who received at least one dose of ranibizumab and had at least one post-baseline safety assessment.
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 7/200
Other Adverse Events (participants affected / at risk) | 26/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=200)
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Klebsiella sepsis (Infections and infestations) | 1
Expired product administered (Study Eye) (Injury, poisoning and procedural complications) | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=200)
Choroidal neovascularisation (Non-study Eye) (Eye disorders) | 3
Choroidal neovascularisation (Study Eye) (Eye disorders) | 7
Conjunctival haemorrhage (Study Eye) (Eye disorders) | 4
Conjunctival hyperaemia (Both Eyes) (Eye disorders) | 5
Ocular hypertension (Both Eyes) (Eye disorders) | 4
Influenza (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.